CLINICAL TRIAL: NCT04449341
Title: Can Virtual Reality Reduce Patient's Pain, Improve Patient's Experience, and Reduce Procedure Related Anxiety With Venipuncture? A Randomized Control Trial
Brief Title: Can Virtual Reality Reduce Pain and Anxiety During Blood Draw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew J. Perdue, DSc, PA-C, Fellow, US Army-Baylor DSc Emergency Medicine PA Studies, Principal Investigator, C.R.Darnall Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 921118
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Procedural Anxiety; Procedural Pain
Keywords: virtual reality; venipuncture; blood draw; Oculus Go
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard care venipuncture with additional of virtual reality (Experimental): Patients undergoing blood draw while interacting with VR application Ocean Rift while wearing Oculus Go headset
  Interventions: Device: Oculus Go headset with Ocean Rift application
- Standard care venipuncture without addition of virtual reality (No Intervention): Patients undergoing blood draw while wearing Oculus Go headset that is turned off

INTERVENTIONS:
Device: Oculus Go headset with Ocean Rift application — Information already included in arm description
  Arms: Standard care venipuncture with additional of virtual reality

SUMMARY:
Adult patients aged 18-50 undergoing blood draw for routine lab evaluation will be randomized to a control group or experimental group to assess if the use of virtual reality reduces procedural pain (primary outcome) and procedural anxiety (secondary outcome) during venipuncture.

DETAILED DESCRIPTION:
A prospective randomized controlled trial comparing standard practice for conducting venipuncture to standard practice with the addition of Virtual Reality using the Oculus Go Head Mounted Display (HMD). The study will be performed on volunteers who are reporting to the phlebotomy lab to have venipuncture for blood draws that were previously ordered by their health care providers. Participants who were not already scheduled to undergo routine venipuncture will not be included.

When approaching the ticket stand to draw a waiting number for the lab, prospective participants will be asked by an assistant investigator located near the kiosk if they are interested in participating in the study. If the participants express interest, they will be directed to the screening station. The screening station will be set up in a private room near the lab waiting area, and participants will be screened for eligibility and educated on the benefits and risks of the study. They will also provide informed consent if they decide to participate.

All participants will be asked to fill out a self-reported data questionnaire in addition to the informed consent document to assess for inclusion and exclusion criteria discussed later in this protocol. This questionnaire will assess the participant's expected level of anxiety prior to the procedure and expected level of pain associated with the procedure by utilizing a visual analog scale (VAS). The VAS will be on a 100 millimeter line.

Once approved for participation in the study all participants will undergo a brief instructional class on how to operate the HMD and will be allowed sufficient time to become comfortable with its use. The investigators expect approximately 5-10 minutes to be required for this portion of the study. Once familiar with the use of the virtual reality headset, participants will be asked to randomly draw an envelope from a container. This envelope will contain a block and sequence number. The block and sequence number will be the subject identification and will correspond to a predetermined number set on a separate document that will determine if the participant will use the HMD during venipuncture or not. The screener will not have immediate access to the list showing which group the participant will be assigned to. One member of the study team will be present in the lab room to ensure the participant uses the virtual reality headset (or not) according to what is randomly drawn. This member of the research team will have the list showing whether or not the participant is assigned to the control arm or the experimental arm. The participants will then proceed to the specimen room to undergo venipuncture.

Venipuncture for both groups will be occur in the non-dominant arm. The reasoning for this is that the Oculus Go requires one free hand to use a controller. This will ensure that the individuals participating are able to effectively use the device. Those unable to undergo venipuncture in the nondominant arm will undergo venipuncture in the dominant arm instead and will use the Oculus Go dominant arm will undergo venipuncture in the dominant arm instead and will use the Oculus Go controller with their non-dominant hand.

Those utilizing the Oculus Go HMD will be interacting with the virtual reality game Ocean Rift. They will utilize a single controller to explore an underwater safari park. Ocean Rift has multiple environments to choose from, including coral reefs, ship wrecks, lagoons, the arctic, and prehistoric seas. Participants may interact with and and learn about different creatures to include dolphins, turtles, orcas, ray, whales, sea lions, manatees, and dinosaurs. During the game users may travel where they please and interact with what they choose. The virtual reality device is equipped with head-tracking software that allows the user to choose direction by looking around. The entire interior and exterior of the headset will be cleaned with alcohol-based wipes after each use. Alcohol will be used since it is generally well-tolerated on human skin, and since it evaporates quickly. The headset will be dried in the open air for a minimum of two minutes between each subject's use.

Those not using the virtual reality will still wear a headset that will simply be turned off. This is to ensure that any significant change noted with the virtual reality is due to the use of virtual reality itself, and not simply due to "blindfolding" the patient during the procedure.

As some patients experiencing anxiety may be tempted to move during the procedure, lab personnel will instruct participants to remain still during venipuncture. Participants will be advised that they may take breaks as needed if anxiety becomes overwhelming.

After undergoing the procedure, each participant will be asked to fill out the postprocedure questionnaire and return it to the study team member present in the lab room, who will clean the headset as the participant completes the questionnaire. This questionnaire assesses the patient's pain intensity and level of anxiety with the VAS similar to the VAS assessing pain, as well as the patient's satisfaction with the visit which will be measured utilizing a Likert scale for individual questions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50
* Currently scheduled to undergo venipuncture

Exclusion Criteria:

* Less than 18 years old or greater than 50 years old
* History of motion sickness (nausea or vertigo)
* Pregnant women
* Reported history of blood borne disease (no request will be made for which disease participant has)
* Use of pain medication(s) on day of study
* Current use of medical devices, including hearing aids, pacemakers, implanted cardiac defibrillators
* Currently experiencing headache/migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Perdue, PA, Principal Investigator — C.R.Darnall Army Medical Center
Locations (1):
- Carl R Darnall Army Medical Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atzori B, Hoffman HG, Vagnoli L, Patterson DR, Alhalabi W, Messeri A, Lauro Grotto R. Virtual Reality Analgesia During Venipuncture in Pediatric Patients With Onco-Hematological Diseases. Front Psychol. 2018 Dec 20;9:2508. doi: 10.3389/fpsyg.2018.02508. eCollection 2018. PMID 30618938
- [Background] Cassidy KL, Reid GJ, McGrath PJ, Finley GA, Smith DJ, Morley C, Szudek EA, Morton B. Watch needle, watch TV: Audiovisual distraction in preschool immunization. Pain Med. 2002 Jun;3(2):108-18. doi: 10.1046/j.1526-4637.2002.02027.x. PMID 15102157
- [Background] Lee JS, Hobden E, Stiell IG, Wells GA. Clinically important change in the visual analog scale after adequate pain control. Acad Emerg Med. 2003 Oct;10(10):1128-30. doi: 10.1111/j.1553-2712.2003.tb00586.x. PMID 14525749
- [Background] Dahlquist LM, Weiss KE, Law EF, Sil S, Herbert LJ, Horn SB, Wohlheiter K, Ackerman CS. Effects of videogame distraction and a virtual reality type head-mounted display helmet on cold pressor pain in young elementary school-aged children. J Pediatr Psychol. 2010 Jul;35(6):617-25. doi: 10.1093/jpepsy/jsp082. Epub 2009 Sep 28. PMID 19786489
- [Background] Garrett B, Taverner T, Masinde W, Gromala D, Shaw C, Negraeff M. A rapid evidence assessment of immersive virtual reality as an adjunct therapy in acute pain management in clinical practice. Clin J Pain. 2014 Dec;30(12):1089-98. doi: 10.1097/AJP.0000000000000064. PMID 24535053
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Gold JI, Belmont KA, Thomas DA. The neurobiology of virtual reality pain attenuation. Cyberpsychol Behav. 2007 Aug;10(4):536-44. doi: 10.1089/cpb.2007.9993. PMID 17711362
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113
- [Background] Hoffman HG, Sharar SR, Coda B, Everett JJ, Ciol M, Richards T, Patterson DR. Manipulating presence influences the magnitude of virtual reality analgesia. Pain. 2004 Sep;111(1-2):162-8. doi: 10.1016/j.pain.2004.06.013. PMID 15327820
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Moore B, Stocks C, Owens P. Trends in Emergency Department Visits, 2006-2014. Healthcare Cost and Utilization Project (HCUP) Statistical Brief #227. 2017
- [Background] Wiederhold BK, Gao K, Kong L, Wiederhold MD. Mobile devices as adjunctive pain management tools. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):385-9. doi: 10.1089/cyber.2014.0202. PMID 24892202
- [Background] Ozalp Gerceker G, Ayar D, Ozdemir EZ, Bektas M. Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1151-1161. doi: 10.1111/jocn.15173. Epub 2020 Jan 22. PMID 31889358
- See also: 2018 Demographics Report: Profile of the Military Community — https://download.militaryonesource.mil/12038/MOS/Reports/2018-demographics-report.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality: Patients undergoing blood draw while interacting with VR application Ocean Rift while wearing Oculus Go headset
  Oculus Go headset with Ocean Rift application: Information already included in arm description
- Control: Patients undergoing blood draw while wearing Oculus Go headset that is turned off
Period: Overall Study
Arm/Group | Virtual Reality | Control
Started | 31 | 28
Completed | 30 | 28
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care Venipuncture With Additional of Virtual Reality | Standard Care Venipuncture Without Addition of Virtual Reality | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 30 | 28 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Procedural Pain
Description: Determine if use of Oculus Go headset reduces procedural pain perception utilizing the visual analog scale, which measures pain on a linear scale from 0 to 100 millimeters, with 0 being no pain and 100 being maximum pain
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Care Venipuncture With Additional of Virtual Reality | Standard Care Venipuncture Without Addition of Virtual Reality
Number analyzed (Participants) | 30 | 28
score on a scale | 6.50 [0.25 to 30.75] | 5.00 [1.00 to 24.25]

2. Secondary Outcome: Procedural Anxiety
Description: Determine if use of Oculus Go headset reduces procedural anxiety utilizing the visual analog scale, which measures anxiety on a linear scale from 0 to 100 millimeters, with 0 being no anxiety and 100 being maximum anxiety
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Care Venipuncture With Additional of Virtual Reality | Standard Care Venipuncture Without Addition of Virtual Reality
Number analyzed (Participants) | 31 | 28
score on a scale | 5 [1.00 to 24.25] | 6.5 [.25 to 30.75]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Standard Care Venipuncture With Additional of Virtual Reality | Standard Care Venipuncture Without Addition of Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04449341/Prot_SAP_000.pdf